CLINICAL TRIAL: NCT01780207
Title: Impact Of Closure Of Patent Foramen Ovale On Apnoea-Hypopnoea-Index, Nocturnal Hypoxemia And Systemic Vascular Function In Patients With Obstructive Sleep Apnoea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Christian Seiler, MD Prof, Insel Gruppe AG, University Hospital Bern
Other Study IDs: 066/10
Record Dates: First submitted 2013-01-29; First posted 2013-01-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

ARMS (2):
- OSA without PFO (No Intervention)
- OSA with PFO (Other): PFO closure
  Interventions: Device: PFO Closure

INTERVENTIONS:
Device: PFO Closure
  Arms: OSA with PFO

SUMMARY:
The purpose of this study in patients with obstructive sleep apnoea (OSA) and concomitant patent foramen ovale (PFO) is to assess the impact of percutaneous PFO closure on nocturnal hypoxemia and apnea/hypopnea, pulmonary and systemic artery pressure, endothelial function and arterial stiffness.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed moderate to severe OSA
* Age > 17 years
* Written informed consent for study participation.

Exclusion Criteria:

* Patients with other pulmonary disease associated with oxygen desaturation (other than obesity-associated pulmonary restriction)
* Patients with central sleep apnea syndrome
* Patients with other causes of pulmonary hypertension
* Intracardiac shunt other than via PFO
* Severe valvular heart disease
* Abnormal left ventricular (LV) systolic function (ejection fraction <50%)
* Obesity with BMI > 40
* Contraindication to TOE
* Severe pulmonary arterial hypertension (mean pulmonary artery pressure > 45 mmHg)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Primary Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Apnea Hypopnea Index (AHI), apnea index (changes from baseline to follow-up) | 0, 3 months

SECONDARY OUTCOMES:
Systemic vascular assessment | 0, 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bern, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Derived] Rimoldi SF, Ott S, Rexhaj E, de Marchi SF, Allemann Y, Gugger M, Scherrer U, Seiler C. Patent Foramen Ovale Closure in Obstructive Sleep Apnea Improves Blood Pressure and Cardiovascular Function. Hypertension. 2015 Nov;66(5):1050-7. doi: 10.1161/HYPERTENSIONAHA.115.06303. Epub 2015 Sep 21. PMID 26418025